CLINICAL TRIAL: NCT02972268
Title: Clinical Trial to Compare the Efficacy and Safety of Solifenacin/Tamsulosin Combination Therapy With Tamsulosin Monotherapy for Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Clinical Trial to Compare the Solifenacin/Tamsulosin Combination Therapy With Tamsulosin Monotherapy for LUTS Due to BPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JLP-1207-P3
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): Tamsulosin 0.2mg + Solifenacin 5mg
  Interventions: Drug: Tamsulosin 0.2mg + Solifenacin 5mg
- Group II (Placebo Comparator): Tamsulosin 0.2mg + Placebo(Solifenacin)
  Interventions: Drug: Tamsulosin 0.2mg + Placebo(Solifenacin)

INTERVENTIONS:
Drug: Tamsulosin 0.2mg + Solifenacin 5mg — Tamsulosin 0.2mg + Solifenacin 5mg for 12wks
  Arms: Group I
Drug: Tamsulosin 0.2mg + Placebo(Solifenacin) — Tamsulosin 0.2mg + Placebo(Solifenacin) for 12wks
  Arms: Group II

SUMMARY:
Clinical Trial to Compare the Efficacy and Safety of Solifenacin/Tamsulosin Combination Therapy with Tamsulosin Monotherapy for Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Over 45 years
* Benign Prostate Hyperplasia diagnosed by 20 mL < TRUS
* Lower urinary tract symptom suggestive of benign prostate hyperplasia, who spontaneously agree to join and sign to the consent form

Exclusion Criteria:

* Subjects who have a history of the lower urinary tract cancer, including prostate cancer and bladder cancer within the past 3 years
* Subjects who have acute urinary retention within 12 weeks before screening
* Subjects who have clinically significant severe cardiovascular disease(unstable angina, myocardial infarction or arrhythmia) within 24 weeks before screening
* Subjects who have hypersensitivity to investigational product
* Subjects who were suspected or confirmed neurogenic bladder, bladder neck structure, bladder diverticulum
* Subjects who have myasthenia gravis, narrow angle glaucoma
* Subjects who have hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* SBP > 180 mmHg or DBP > 100 mmHg
* HbA1c > 9.0 %
* Subjects who are judged by the investigators to be unsuitable to participate in the clinical trial.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
change of TUFS | 12 weeks from baseline
change of total IPSS | 12 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Myung Soo Choo, MD., Ph.D, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No